CLINICAL TRIAL: NCT06131372
Title: Efficacy and Safety of Co-administered Cagrilintide and Semaglutide (CagriSema 2.4 mg/2.4 mg) Once Weekly Versus Semaglutide 2.4 mg, Cagrilintide 2.4 mg and Placebo in People With Chronic Kidney Disease and Type 2 Diabetes Living With Overweight or Obesity
Brief Title: A Research Study to See if Kidney Damage in People With Chronic Kidney Disease and Type 2 Diabetes Living With Overweight or Obesity Can be Reduced by CagriSema Compared to Semaglutide, Cagrilintide and Placebo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-7700; U1111-1291-5907 (Other: World Health Organization (WHO)); 2023-505857-42 (EudraCT Number)
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes; Obesity
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2; Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CagriSema (Experimental): Participants will receive cagrilintide and semaglutide subcutaneously once-weekly after a dose escalation period of 16 weeks during the maintenance period for 10 weeks.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide
- Semaglutide (Experimental): Participants will receive semaglutide and placebo matched to cagrilintide subcutaneously once-weekly after a dose escalation period of 16 weeks during the maintenance period for 10 weeks.
  Interventions: Drug: Semaglutide; Drug: Placebo
- Cagrilintide (Experimental): Participants will receive cagrilintide and placebo matching to semaglutide subcutaneously once-weekly after a dose escalation period of 16 weeks during the maintenance period for 10 weeks.
  Interventions: Drug: Cagrilintide; Drug: Placebo
- Placebo (Placebo Comparator): Participants will receive placebo matched to cagrilintide and placebo matched to semaglutide subcutaneously once weekly for 26 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive Cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide
Drug: Semaglutide — Participants will receive semaglutide subcutaneously.
  Arms: CagriSema; Semaglutide
Drug: Placebo — Participants will receive placebo matched to cagrilintide or placebo matched to semaglutide subcutaneously.
  Arms: Cagrilintide; Placebo; Semaglutide

SUMMARY:
This study will look if CagriSema can lower kidney damage in people with chronic kidney disease (CKD), type 2 diabetes (T2D) and overweight or obesity. CagriSema is a new investigational medicine. CagriSema cannot yet be prescribed by doctors. The study will compare CagriSema to the 2 medicines semaglutide and cagrilintide, when they are taken alone. It will also compare CagriSema to a "dummy" medicine (also called placebo) without any active ingredient. Participant will either get CagriSema, semaglutide, cagrilintide or placebo. Which treatment participant will get is decided by chance (like flipping a coin). Study doctor will not know which of the study medicines participant will get. For each participant, the study will last for about 35 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female.
* Age 18 years or above at the time of signing the informed consent.
* Diagnosed with type 2 diabetes mellitus ≥ 180 days before screening.
* Body mass index (BMI) ≥ 27.0 kilograms per meter square (kg/m^2) at screening. BMI will be calculated in the eCRF (electronic case report form) based on height and body weight at screening.
* HbA1c less than or equal to (≤) 10.5% (91 millimoles per mole [mmol/mol]) as assessed by central laboratory at screening.
* Kidney impairment defined by serum creatinine and cystatin C-based eGFR ≥ 15 and < 90 milliliters per minutes per 1.73^m^2 (mL/min/1.73 m^2) (CKD-EPI 2021) as assessed by central laboratory at screening.
* Albuminuria defined by UACR ≥ 100 and < 5000 milligram per gram (mg/g) as assessed by central laboratory at screening.
* Treatment with maximum labelled or tolerated dose of an angiotensin converting enzyme (ACE) inhibitor or an angiotensin II receptor blocker (ARB), unless such treatment is contraindicated or not tolerated, in the opinion of the investigator. Treatment dose must be stable for at least 30 days prior to screening.

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using a highly effective contraceptive method.
* Congenital or hereditary kidney diseases including polycystic kidney disease, autoimmune kidney diseases including glomerulonephritis or congenital urinary tract malformations.
* Use of any glucagon-like peptide-1 receptor agonist (GLP-1RA) (including medication with GLP-1RA activity, e.g., GIP/GLP-1RA) or amylin analogue within 60 days prior to screening.
* Myocardial infarction, stroke, transient ischaemic attack, or hospitalization for unstable angina pectoris within 60 days before screening.
* Chronic or intermittent haemodialysis or peritoneal dialysis within 90 days before screening.
* Uncontrolled and potentially unstable diabetic retinopathy or maculopathy. Verified by an eye examination performed within 90 days before screening or in the period between screening and randomisation. Pharmacological pupil-dilation is a requirement unless using a digital fundus photography camera specified for non-dilated examination.
* Presence or history of malignant neoplasms or in situ carcinomas (other than basal or squamous cell skin cancer, low-risk prostate cancer, or in-situ carcinomas of the cervix or carcinoma in situ/high grade prostatic intraepithelial neoplasia (PIN) within 5 years before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-09-24 (Actual); Study Completion 2025-11-06 (Actual)

PRIMARY OUTCOMES:
Change in urinary albumin-to-creatinine ratio (UACR) | From baseline (week 0) to end of treatment (week 26)
  Measured in ratio to baseline.

SECONDARY OUTCOMES:
Change in estimated glomerular filtration rate (eGFR) (creatinine and cystatin C-based chronic kidney disease (CKD)-Epidemiology Collaboration equation (EPI) 2021) | From baseline (week 0) to end of treatment (week 26)
  Measured in milliliters per minute per 1.73 meters square (mL/min/1.73 m^2).
Change in eGFR (creatinine-based CKD-EPI 2021) | From baseline (week 0) to end of treatment (week 26)
  Measured in mL/min/1.73 m^2.
Relative change in body weight | From baseline (week 0) to end of treatment (week 26)
  Measured in percentage (%).
Achievement of greater than or equal to (≥) 5 % weight reduction | From baseline (week 0) to end of treatment (week 26)
  Count of participants.
Achievement of ≥ 10 % weight reduction | From baseline (week 0) to end of treatment (week 26)
  Count of participants.
Change in waist circumference | From baseline (week 0) to end of treatment (week 26)
  Measured in centimeter (cm).
Change in glycated haemoglobin (HbA1c) | From baseline (week 0) to end of treatment (week 26)
  Measured in %-points.
Change in systolic blood pressure | From baseline (week 0) to end of treatment (week 26)
  Measured in millimeters of mercury (mmHg).
Change in diastolic blood pressure | From baseline (week 0) to end of treatment (week 26)
  Measured in mmHg.
Number of treatment emergent adverse events (TEAEs) | From baseline (week 0) to end of study (week 32)
  count of events.
Number of treatment emergent serious adverse events (SAEs) | From baseline (week 0) to end of study (week 32)
  count of events.
Number of clinically significant hypoglycaemic episodes (level 2) ( blood glucose less than [<] 3.0 millimoles per liter [mmol/L] (54 milligram per deciliter [mg/dL])) | From baseline (week 0) to end of study (week 32)
  Count of episodes.
Number of severe hypoglycaemic episodes (level 3): hypoglycaemia associated with severe cognitive impairment requiring external assistance for recovery, with no specific glucose threshold | From baseline (week 0) to end of study (week 32)
  Count of episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (122):
- United States (25):
  - John Muir Physicians Network, Concord, California
  - Valley Research, Fresno, California
  - Desert Oasis Hlthcr Med Group, Palm Springs, California
  - North America Research Institute, San Dimas, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Northeast Research Institute, Fleming Island, Florida
  - Life Spring Research, Miami, Florida
  - Florida Hospital Translational Research Institute, Orlando, Florida
  - Velocity Clin. Res Valparaiso, Valparaiso, Indiana
  - Elite Research Center, Flint, Michigan
  - Univ. of Nebraska Medical Center_Omaha, Omaha, Nebraska
  - Albany Medical College, Albany, New York
  - NYU Langone Neph Associates, Mineola, New York
  - New York University School of Medicine, New York, New York
  - Southgate Medical Group, LLP, West Seneca, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Eastern Nephr Assoc, PLLC, New Bern, North Carolina
  - Brookview Hills Research Associates, LLC, Winston-Salem, North Carolina
  - Ohio- Advanced Medical Research, Maumee, Ohio
  - Heritage Valley Medical Group Inc, Beaver, Pennsylvania
  - Main Street Physician's Care, Little River, South Carolina
  - Osvaldo A. Brusco MD PA, Corpus Christi, Texas
  - Southwest Houston Research Ltd, Houston, Texas
  - Clinical Advancement Ctr, PLLC, San Antonio, Texas
  - Clinical Investigation Spec. Kenosha, Kenosha, Wisconsin
- Argentina (5):
  - Mautalen Salud e investigación, CABA, Buenos Aires
  - Centro de Investigaciones Médicas Mar del Plata, Mar del Plata, Buenos Aires
  - Fundación CESIM, Santa Rosa, La Pampa Province
  - Centro Medico Dra. Laura Maffei e Investigacion Clínica Apli, Buenos Aires
  - Centro Médico Privado San Vicente Diabetes, Córdoba
- Brazil (4):
  - Instituto Pró-Renal Brasil, Curitiba, Paraná
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul Ltda., Porto Alegre, Rio Grande do Sul
  - CPCLIN - Centro de Pesquisas Clínicas, São Paulo, São Paulo
  - Hospital do Rim e Hipertensao Fundacao Oswaldo Ramos, São Paulo
- Canada (9):
  - Centricity Research Calgary, Calgary, Alberta
  - Centricity Research Brampton, Brampton, Ontario
  - Centricity Research Vaughn Endocrinology, Concord, Ontario
  - Centricity Research Etobicoke, Etobicoke, Ontario
  - Hamilton Medical Rsrch Grp, Hamilton, Ontario
  - Bluewater Clin Res Group Inc, Sarnia, Ontario
  - UHN-Toronto General Hospital, Toronto, Ontario
  - Ctr de rech Clin de Laval, Laval, Quebec
  - Centre Medical Acadie, Montreal, Quebec
- France (7):
  - Groupe Sos Sante-Hopital Le Creusot-Hotel Dieu-1, Le Creusot
  - Gie Groupe Hospitalier Paris Saint-Joseph/Vinci, Paris
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Centre Hospitalier Universitaire Reims-Hopital Maison Blanche, Reims
  - Centre Hospitalier Universitaire de Nantes-Hopital Nord Laennec-1, Saint-Herblain
  - Centre Hospitalier Universitaire de Toulouse-Hopital Rangueil-1, Toulouse
  - Centre de Recherche Clinique Portes Du Sud, Vénissieux
- Greece (14):
  - University General Hospital Of Heraklion, Heraklion, Crete
  - "Laiko" General Hospital of Athens, Athens
  - Gen Hospital of Athens Laiko,1st Dpt. of Propaedeutic Inter, Athens
  - General hospital of Athens 'G.Gennimatas', Athens
  - Iatriko Athinon 'Palaiou Falirou', Athens
  - General Hospital of Lamia, Lamia
  - Univ Gen Hospital Larisa, Larissa
  - Univ Gen Hospital Larisa, Endocrinology & Metabolic Disease, Larissa
  - General University Hospital of Patras,Nephrology clinic, Pátrai
  - General University Hospital of Patras,Nephrology clinic, Rio, Patra
  - General Hospital of Thessaloniki 'G. Gennimatas, Thessaloniki
  - "Ippokrateio" G.H. of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "Ippokrateio", Thessaloniki
  - General Hospital of Thessaloniki "G.Papanikolaou", Thessaloniki
- Hungary (7):
  - PTE-AOK II. Belgyogyaszati Klinika es Nephrologiai Centrum, Pécs, Baranya Vármegye
  - Lausmed Kft., Baja, Bács-Kiskun county
  - Belinus Bt., Debrecen, Hajdú-Bihar
  - Siófoki Kórház, Diabetológiai Szakrendelés, Siófok, Somogy County
  - Borbánya Praxis E.Ü. Kft., Nyíregyháza, Szabolcs-Szatmar Varmegye
  - Szent Margit Rendelőintézet Nonprofit Kft., Budapest
  - Békés Megyei Központi Kórház, Gyula
- India (9):
  - Endolife Specialty Hospitals, Guntur, Andhra Pradesh
  - NIZAM'S Institute of Medical Sciences, Hyderabad, Andhra Pradesh
  - Sunrise Hospital, Vijayawada, Andhra Pradesh
  - Lifecare Hospital and Research Centre, Bengaluru, Karnataka
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - King Edward Memorial Hospital, Pune- Maharashtra, Maharashtra
  - Maulana Azad Medical College, Delhi, New Delhi
  - Madras Diabetes Research Foundation, Chennai, Tamil Nadu
  - Shri Mahant Indiresh Hospital, Dehradun, Uttarakhand
- Japan (9):
  - Seino Internal Medicine Clinic_Internal medicine, Koriyama-shi, Fukushima, Japan
  - Nippon Kokan Fukuyama Hospital_Diabetology, Fukuyama-shi, Hiroshima
  - Sasaki Internal Medicine, Hokkaido
  - Nishiyamado Keiwa Hospital_Internal Medicine, Ibaraki
  - Kanno Naika_Internal Medicine, Mitaka-shi, Tokyo
  - Minami Akatsuka Clinic, Mito-shi, Ibaraki
  - Tokyo-Eki Center-building Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic_Internal Medicine, Tokyo
  - Fukuwa Clinic, Tokyo
- Poland (13):
  - Osteo Medic s.c. Artur Racewicz Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - NZOZ Specjalistyczny Osrodek Internistyczno-Diabetologiczny Małgorzata Arciszewska, Bialystok, Podlaskie Voivodeship
  - Kresmed Sp. z o. o., Bialystok, Podlaskie Voivodeship
  - M2M Med. Sp. z o.o. Sp. j., Chorzów, Silesian Voivodeship
  - M2M Med. Sp. z o.o. Sp. j., Chorzów
  - Pratia S.A., Gdynia
  - Pratia S.A., Katowice
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz
  - Etyka Osrodek Badan Klinicznych Tomasz Pesta S.K.A., Olsztyn
  - Gaja Poradnie Lekarskie, Poznan
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych I Administracji, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 im. Prof. Szyszko, Zabrze
- Slovakia (6):
  - KARDIO-SANUS, spol. s r.o., Bratislava
  - MEDISPEKTRUM s.r.o., Bratislava
  - HUMAN-CARE, s.r.o., Košice
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Vysokospecializovany odborny ustav geriatricky sv. Lukasa v Kosiciach, n.o., Košice
  - Tatratrial s.r.o., Rožňava
- Spain (7):
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital Fundación Alcorcón, Alcorcón
  - Hospital Vall d'Hebron, Barcelona
  - Hospital de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Gregorio Marañón, Madrid
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Clinico Universitario de Valencia, Valencia
- Thailand (7):
  - Siriraj Hospital, Bangkok Noi, Bangkok
  - Thammasat Hospital, Klong Luang Pathum Thani, Changwat Pathum Thani
  - Thammasat University Hospital, Klong Luang, Changwat Pathum Thani
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai, Mueang Chiang Mai
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com